CLINICAL TRIAL: NCT03079986
Title: Chyle Leak After Pancreatic Surgery - CLAP
Brief Title: Chyle Leak After Pancreatic Surgery
Acronym: CLAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Jan D'Haese, Associate professor, principal investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAP
Record Dates: First submitted 2017-02-25; First posted 2017-03-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Chyle Leak
Keywords: Pancreatic surgery; Chylous ascites
MeSH Terms: conditions — Chylous Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ignoring CL (group A) (Experimental): Standard care irrespective of CL.
  Interventions: Other: Standard care irrespective of CL
- Dietary treatment (group B) (Active Comparator): Dietary treatment with medium-chain triglyceride diet (MCT-diet) until resolution of CL.
  Interventions: Other: Dietary treatment (MCT-diet)

INTERVENTIONS:
Other: Standard care irrespective of CL — Removal of surgical drains despite persistent CL, without dietary restrictions or dietary treatment for CL.
  Arms: Ignoring CL (group A)
Other: Dietary treatment (MCT-diet) — Dietary treatment with MCT-diet until resolution of CL.
  Arms: Dietary treatment (group B)

SUMMARY:
Currently it is unclear whether postoperative chyle leak (CL) after pancreatic surgery requires treatment. Thus, the present study aims to compare dietary treatment of CL with drain removal despite of persistent CL.

DETAILED DESCRIPTION:
With an incidence of up to 11%, postoperative chyle leak (CL) is a frequent phenomenon after pancreatic surgery, where extensive lymph node dissections are indispensable. Postoperative CL is frequently treated with either medium-chain triglyceride diet (MCT-diet) or total parenteral nutrition (TPN). Ignoring CL and removing the surgical drains irrespective of CL may also be discussed. While dietary restrictions are known to hinder postoperative convalescence and prolong the length of stay at the hospital, recent retrospective data show that leaving CL untreated is not associated with an increased morbidity rate. More precisely, removing the surgical drains irrespective of CL does not result in an increased incidence of CT-guided drainages. However, prospective data on CL after pancreatic surgery do not exist in the literature. Accordingly, the present trial aims to compare treatment of CL with dietary restrictions to removing the surgical drains irrespective of CL.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Pancreatic surgery of any kind

Exclusion Criteria:

* Liver cirrhosis > Child-Pugh grade A
* History of portal vein thrombosis
* Portal Hypertension

Dropout Criteria:

* Irresectable Tumor (no surgical resection)
* Biochemical leak or postoperative pancreatic fistula (POPF)5
* Serous drainage on POD 5
* Peritoneal carcinomatosis
* Portal vein thrombosis
* Postoperative bile leak
* Drain volume >1000ml on POD5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative morbidity | 30 days postoperatively
  Complications ≥ Clavien-Dindo3 grade IIIa

SECONDARY OUTCOMES:
Length of stay at the hospital | 90 days postoperatively
  The time spent at the hospital will be recorded
Time until drain removal | 30 days postoperatively
  The time until drain removal will be recorded
Readmission to the hospital | 90 days postoperatively
  Patients will be called and asked for any readmission to a hospital (yes /no)
Weight change | The day before surgery until postoperative day 10
  Weight (Day before surgery) - Weight (10 days postoperatively)
Body mass index (BMI) change | The day before surgery until postoperative day 10
  BMI (day before surgery) - BMI (10 days postoperatively)
International normalized ration (INR) change | The day before surgery until postoperative day 10
  INR (Day before surgery) - INR (10 days postoperatively)
Albumin change | The day before surgery until postoperative day 10
  Albumin level (Day before surgery) - Albumin level (10 days postoperatively)
Postoperative cortisol level | 8 days postoperatively
  Cortisol levels will be compared between group A and B
Freiburg index of patient satisfaction | Postoperative day 10
  Patient satisfaction will be measured using a standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jan D'Haese, M.D., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Ludwig-Maximilians-University, Munich, Germany